CLINICAL TRIAL: NCT05291429
Title: Study to Identify if OVR Health's VR-Kit is Safe to Use and Helps Individuals to Improve Focus, Attention and Reduce Worry & Rumination.
Brief Title: Study to Identify if OVR Health's VR-Kit is Safe to Use and Helps to Improve Focus, Attention and Reduce Worry & Rumination.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford VR (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20213Oxford
Record Dates: First submitted 2022-01-31; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Anxiety; Depression, Anxiety
Keywords: Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR - coaching arm (Active Comparator): 30 individuals to be enrolled in the intervention arm that also includes coaching sessions to support and encourage VR use (VR+coaching arm).
  Interventions: Device: OVR Health's VR experience
- VR only - no coaching (Active Comparator): 30 individuals to be enrolled in the intervention arm without coaching (VR arm)
  Interventions: Device: OVR Health's VR experience
- No intervention - control arm (No Intervention): 30 individuals to be enrolled in the control arm with no active intervention (comparator 2; control arm)

INTERVENTIONS:
Device: OVR Health's VR experience — Virtual reality experience
  Arms: VR - coaching arm; VR only - no coaching

SUMMARY:
This is a randomized-controlled interventional treatment study with three arms of comparable demographics to evaluate the safety and efficacy of OVR Health's VR experience to improve control over the focus of attention and reduce worry and rumination in individuals who have reported problems with these issues.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Must be in good general health
* Self-reported with the following symptoms (as assessed by questions and questionnaires in study material):
* Finding it hard to let go of difficult thoughts.
* Looking out for signs of a potential threat in their environment (or in their body) that unhelpfully maintains their problem.
* Engaging in repetitive, unhelpful patterns of negative thinking (worry & rumination). • These may be due to a diagnosis of a mental health condition, but this is not required for entry into the study.
* Good understanding of written and spoken English
* Willing and able to give informed consent
* Willing and able to follow the study protocol
* Willing and able to use VR headset at home
* WiFi connection to connect VR headset at home
* Willing and able to return VR headset

Exclusion Criteria:

* Current diagnosis of epilepsy, dementia, or another neurological disease that may prevent the use of VR hardware and software
* Individuals with suicidal or self-harm thoughts
* Significant visual, auditory, or balance impairment
* Insufficient comprehension of English
* Primary diagnosis of alcohol or substance abuse disorder, or personality disorder • Significant learning disability
* Current active suicidal plans or self-harm (in which case participant will be referred to appropriate crisis service)
* Receiving current alternative psychotherapy treatment
* Unwilling to provide consent
* Unwilling to follow the study protocol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Safety of virtual reality device and reduction in worry and rumination (PHQ9) | 5 weeks
  Changes in perceived safety using the PHQ9 questionnaire (Scale 0-3).
Safety of virtual reality device and reduction in worry and rumination (Perseverative Thinking score ) | 5 weeks
  Changes in perceived safety using the Perseverative Thinking score (Scale 0-4).

SECONDARY OUTCOMES:
Impact of coaching on virtual reality intervention effectiveness (PHQ9) | 5 weeks
  Changes in the PHQ9 questionnaire (0-3) in comparison to Group 2 (no coaching) and placebo arm (no intervention) with a lower score showing fewer symptoms.
Impact of coaching on virtual reality intervention effectiveness (Perseverative Thinking scor) | 5 weeks
  Changes in the Perseverative Thinking score (0-4) in comparison to Group 2 (no coaching) and placebo arm (no intervention) with a lower score showing fewer symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No